CLINICAL TRIAL: NCT07118176
Title: PET Imaging Study of 68Ga-FAPI-46 Biodistribution in Cancer Patients
Brief Title: Determining the Biodistribution of an Imaging Tracer (68Ga-FAPi-46) in Patients With Solid Tumors or Hematologic Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-0201; NCI-2025-04961 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Anal Carcinoma; Bladder Carcinoma; Breast Carcinoma; Cervical Carcinoma; Cholangiocarcinoma; Colorectal Carcinoma; Esophageal Carcinoma; Gastric Carcinoma; Head and Neck Carcinoma; Hematopoietic and Lymphatic System Neoplasm; Hepatocellular Carcinoma; Lung Carcinoma; Malignant Adrenal Gland Neoplasm; Malignant Brain Neoplasm; Malignant Neoplasm of Unknown Primary; Malignant Solid Neoplasm; Malignant Testicular Neoplasm; Malignant Uterine Neoplasm; Neuroendocrine Neoplasm; Ovarian Carcinoma; Pancreatic Carcinoma; Penile Carcinoma; Pleural Carcinomatosis; Primary Peritoneal Carcinoma; Prostate Carcinoma; Salivary Gland Carcinoma; Sarcoma; Skin Carcinoma; Solitary Fibrous Tumor; Thymus Carcinoma; Thyroid Gland Carcinoma; Thyroid Gland Medullary Carcinoma; Urothelial Carcinoma; Vaginal Carcinoma
MeSH Terms: conditions — Anus Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Cholangiocarcinoma; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Adrenal Gland Neoplasms; Brain Neoplasms; Testicular Neoplasms; Uterine Neoplasms; Neuroendocrine Tumors; Ovarian Neoplasms; Pancreatic Neoplasms; Penile Neoplasms; Prostatic Neoplasms; Salivary Gland Neoplasms; Sarcoma; Solitary Fibrous Tumors; Thyroid Neoplasms; Carcinoma, Medullary; Carcinoma, Transitional Cell; Vaginal Neoplasms | interventions — Fluorodeoxyglucose F18; FAPI-46; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (68Ga-FAPi-46 PET/CT) (Experimental): Patients receive 68Ga-FAPi-46 IV and then, 20-90 minutes later, undergo PET/CT over 20-50 minutes. Patients may undergo optional 18F-FDG PET/CT on study.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Radiation: Gallium Ga 68 FAPi-46; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: Gallium Ga 68 FAPi-46 — Given IV
  Other Names: (68GA)Ga-FAPI-46; 68Ga-FAPi-46; FAPI-46 GA-68; Gallium-68-FAPI-46
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial is evaluating a new imaging tracer (68Ga-FAPi-46) with positron emission tomography (PET)/computed tomography (CT) to determine where and to which degree the tracer (68Ga-FAPi-46) accumulates in normal and cancer tissues (the biodistribution) in patients with solid tumors or hematologic (blood) cancers. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, 68Ga-FAPi-46. Because some cancers take up 68Ga-FAPi-46, it can be seen with PET. CT utilizes x-rays that traverse the body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in a patient's body. Combining a PET scan with a CT scan can help make the image easier to interpret. PET/CT scans are hybrid scanners that combine both modalities into a single scan during the same examination.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the biodistribution of gallium Ga 68 FAPi-46 (68Ga-FAPi-46) in normal and cancer tissues of patients with various malignancies measured by standardized uptake values (SUV).

SECONDARY OBJECTIVE:

I. To assess the 68Ga-FAPI-46 biodistribution correlation with fludeoxyglucose F-18 (18F-FDG) biodistribution and to define the frequency of the following phenotypes (FAP+/ FDG+, FAP-/ FDG+, FAP+/ FDG-, FAP-/ FDG-).

OUTLINE:

Patients receive 68Ga-FAPi-46 intravenously (IV) and then, 20-90 minutes later, undergo PET/CT over 20-50 minutes. Patients may undergo optional 18F-FDG PET/CT on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following suspected or diagnosed cancer types:

  * Adrenal cancer
  * Anal cancer
  * Bladder cancer
  * Brain cancer
  * Breast cancer
  * Cancer of unknown primary (CUP)
  * Cervical cancer
  * Cholangiocarcinoma
  * Colorectal cancer
  * Esophageal cancer
  * Gastric cancer
  * Head and neck cancer
  * Hematologic cancer
  * Hepatocellular carcinoma
  * Lung cancer
  * Medullary thyroid cancer
  * Neuroendocrine neoplasias
  * Ovarian cancer
  * Pancreatic cancer
  * Penile cancer
  * Peritoneal cancer
  * Pleural cancer
  * Prostate cancer
  * Sarcoma
  * Salivary gland cancer
  * Solitary fibrous tumor
  * Skin cancer
  * Testicular cancer
  * Thymus cancer
  * Thyroid cancer
  * Urothelial cancer
  * Uterus cancer
  * Vaginal cancer
* Patients are ≥ 18 years old at the time of the radiotracer administration
* Patient can provide written informed consent
* Patient is able to remain still for duration of imaging procedure (up to one hour)

Exclusion Criteria:

* Patient is pregnant or nursing
* Patient has underlying disease which, based on the judgment of the investigator, might interfere with the collection of high-quality data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2027-09-07 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of gallium Ga 68 FAPi-46 (68Ga-FAPi-46) | Up to 2 years
  Will be evaluated in normal and cancer tissues by standardized uptake values to determine where and to which degree 68Ga-FAPi-46 accumulates in normal and cancer tissues.

SECONDARY OUTCOMES:
Fludeoxyglucose F-18 (18F-FDG) biodistribution | Up to 2 years
  Will assess the correlation between 68Ga-FAPi-46 biodistribution and 18F-FDG biodistribution and define the frequency of the following phenotypes: 68Ga-FAPi-46 (FAP)+/fludeoxyglucose F-18 (FDG)+, FAP-/FDG+, FAP+/FDG-, FAP-/FDG-.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States